CLINICAL TRIAL: NCT05067764
Title: Multicenter, Randomized, Open-label Study Evaluating the Efficacy of Aponeurectomy Associated With Adipose Tissue Grafting Compared to Aponeurectomy Alone, on the 2-year Recurrence Rate of Dupuytren's Disease (REMEDY).
Brief Title: Efficacy of Aponeurectomy on the 2-year Recurrence Rate of Dupuytren's Disease
Acronym: REMEDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REMEDY; 2020-A03214-35 (Other: ANSM)
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, therapeutic, comparative, randomized controlled open-label, superiority, multicenter, national study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aponeurectomy with grafting (Experimental): The experimental group evaluates the aponeurectomy associated with adipose tissue grafting.
  Interventions: Procedure: Aponeurectomy with grafting
- Aponeurectomy alone (Active Comparator): The control group evaluates the aponeurectomy alone.
  Interventions: Procedure: Aponeurectomy alone

INTERVENTIONS:
Procedure: Aponeurectomy with grafting — The lipofilling is performed, once the incisions are closed and is performed with the Puregraft® system.
  The fat graft is taken from the posterior, medial and anterior sides of the arm, by skin puncture. Approximately 10 cc are harvested, allowing a reinjection of about 2 cc per digital radius treated. After conditioning, the fat graft is redistributed to the curettage areas through the skin incisions.
  Arms: Aponeurectomy with grafting
Procedure: Aponeurectomy alone — The patient is installed in dorsal decubitus position and the arm to be treated is anesthetized by axillary block. The procedure is performed in the operating room, respecting all the rules of asepsis and safety in force. A tourniquet is placed on the arm to be treated and inflated to 250mmHg. Broken incisions are then made opposite the cords to be excised, which are located by palpation. Once the noble elements have been identified, the excision of the cords and fibrous nodules can be done as completely as possible. Sometimes an arthrolysis procedure is necessary in order to restore extension to a joint that has been fixed in a flexion position for several years. Skin closure is most often possible by direct suture or by means of local fatty skin flaps. In some cases, the surgeon may use total skin grafts, or directed healing in certain areas where direct skin suture is not possible.
  Arms: Aponeurectomy alone

SUMMARY:
Dupuytren's disease is a frequent hereditary disease in Northern Europe. It is a degenerative disease affecting the palmar aponeurosis of the hand. It develops a progressive contractile fibrosis which cuts the hypodermic fatty tissue, adheres to the skin and the phalanges, gradually bending the affected rays, resulting in significant functional impotence.

Various medical and surgical treatments are available.

DETAILED DESCRIPTION:
Among these treatments, none to date can eliminate recurrences, which are still too frequent.

Open aponeurectomy (consisting of surgical curettage of the fibrotic cords) remains for the moment the reference technique for treating Dupuytren's disease, with recurrences (between 12 and 39%), but less frequent than the needle technique (50 to 85%).

Could the addition of adipose tissue in the resection areas of Dupytren's fibrosis reduce the rate of recurrence (by the inhibitory action of ADCs on myofibroblasts) in addition to reconstructing the hypodermis in the cavity left by the resection of the cords and improving the quality of the scars? The investigators insist on the fact that this is a homotopic and homologous adipose tissue graft, in closed circuit without denaturation or adjuvant products.

Since, to our knowledge, no other team has used "lipofilling" as an adjuvant treatment to the open resection technique of Dupuytren's cords (aponeurectomy), the investigators first conducted a clinical feasibility and safety study on 70 patients between 2012 and 2017 (currently being published by Springer Editions).

The investigators now wish to conduct a prospective comparative study between patients operated by aponeurectomy WITH (experimental group) and WITHOUT (control group) addition of autologous adipose tissue in the resection areas of Dupuytren's cords.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Carrier of Tubiana stage II-IV Dupuytren's disease on at least one or more rays, not previously operated
* Indication of a surgery by aponeurectomy
* Skin pinch of the posterior aspect of the arm of more than 1cm
* Affiliation to a social security system
* Patient informed of the study and having given informed consent

Exclusion Criteria:

* Previous surgery of any kind for Dupuytren's disease
* Involvement on the thumb only
* Need for a total skin graft or a pedicle flap on all the rays to be treated
* Active autoimmune disease
* Previous treatment with collagenase
* Pregnant and breastfeeding women
* Patient under legal protection
* Contraindications to MRI (criteria applicable only for patients from the coordinating center, not applicable for other centers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2029-09-29 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence rate of Dupuytren's disease | 2 Years after intervention
  Recurrence being defined as follows: appearance, at 2 years post-op compared to 6 weeks post-op, of a contracture of more than 20 degrees, with palpable cord, on any treated joint.

SECONDARY OUTCOMES:
3-year recurrence rate in both groups | 3 Years after intervention
  Recurrence being defined as follows: Appearance of a contracture of more than 20 degrees, with palpable cord, on any treated joint, at 3 years post-op compared to 6 weeks post-op
5-year recurrence rate in both groups | 5 Years after intervention
  Recurrence being defined as follows: Appearance of a contracture of more than 20 degrees, with palpable cord, on any treated joint, at 5 years post-op compared to 6 weeks post-op
Comparison of the appearance of scars in both groups | 1 Year after intervention
  Use of questionnaire The Patient and Observer Scar Assessment Scale (POSAS). This questionnaire consists of 2 separate scales of 6 items each (one scale for the observer and one scale for the patient). Each item is evaluated on 10 points. The lowest score is "1" which corresponds to the appearance of normal skin. A score of 10 indicates the greatest deviation from normal skin. The total score for each of the scales is obtained by adding the score for each of the 6 items. This total score can vary between 6 and 60 for each of the scales.
Comparison of the appearance of scars in both groups | 2 Years after intervention
  Use of questionnaire The Patient and Observer Scar Assessment Scale (POSAS). This questionnaire consists of 2 separate scales of 6 items each (one scale for the observer and one scale for the patient). Each item is evaluated on 10 points. The lowest score is "1" which corresponds to the appearance of normal skin. A score of 10 indicates the greatest deviation from normal skin. The total score for each of the scales is obtained by adding the score for each of the 6 items. This total score can vary between 6 and 60 for each of the scales.
Comparison of the complication rates in both groups | 1 Week after intervention
  Complications are defined as Hematoma, infection, graft lysis, disunion or nerve damage.
Comparison of the complication rates in both groups | 6 Weeks after intervention
  Complications are defined as Hematoma, infection, graft lysis, disunion or nerve damage.
Comparison of the rate of occurrence of algodystrophy, regardless of cause | 1 Year after intervention
  Collection of information on the occurrence of algodystrophy, considered as Adverse Event of Special Interest.
Comparison of the rate of occurrence of algodystrophy, regardless of cause | 2 Years after intervention
  Collection of information on the occurrence of algodystrophy, considered as Adverse Event of Special Interest.
Comparison of the rate of occurrence of algodystrophy, regardless of cause | 3 Years after intervention
  Collection of information on the occurrence of algodystrophy, considered as Adverse Event of Special Interest.
Comparison of the rate of occurrence of algodystrophy, regardless of cause | 5 Years after intervention
  Collection of information on the occurrence of algodystrophy, considered as Adverse Event of Special Interest.
Comparison of the effect on quality of life in both groups | 6 Weeks after intervention
  Use of Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. The score consists of 11 questions that assess the function of the upper limb for the gestures of daily life. The final score is between 0 and 100, with 0 corresponding to normal function, and 100 to almost no function.
Comparison of the effect on quality of life in both groups | 1 Year after intervention
  Use of Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. The score consists of 11 questions that assess the function of the upper limb for the gestures of daily life. The final score is between 0 and 100, with 0 corresponding to normal function, and 100 to almost no function.
Comparison of the effect on quality of life in both groups | 2 Years after intervention
  Use of Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. The score consists of 11 questions that assess the function of the upper limb for the gestures of daily life. The final score is between 0 and 100, with 0 corresponding to normal function, and 100 to almost no function.
Comparison of the effect on quality of life in both groups | 5 Years after intervention
  Use of Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. The score consists of 11 questions that assess the function of the upper limb for the gestures of daily life. The final score is between 0 and 100, with 0 corresponding to normal function, and 100 to almost no function.
Evaluation of the primary endpoint on the second hand operated on. | Within five years after intervention
  The surgery being done with or without fat according to the treatment of the 1st randomized hand (cross-over scheme).
  Data collection for the second surgery only if it occurs between the 1st hand surgery and the patient's protocol discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Elias SAWAYA, MD, Principal Investigator — Institut Aquitain de la Main
Locations (2):
- France (2):
  - Institut Aquitain de la Main, Pessac
  - Santé Atlantique ELSAN, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selles RW, Zhou C, Kan HJ, Wouters RM, van Nieuwenhoven CA, Hovius SER. Percutaneous Aponeurotomy and Lipofilling versus Limited Fasciectomy for Dupuytren's Contracture: 5-Year Results from a Randomized Clinical Trial. Plast Reconstr Surg. 2018 Dec;142(6):1523-1531. doi: 10.1097/PRS.0000000000004982. PMID 30489526
- [Background] Henry M. Dupuytren's disease: current state of the art. Hand (N Y). 2014 Mar;9(1):1-8. doi: 10.1007/s11552-013-9563-0. PMID 24570630
- [Background] Engstrand C, Krevers B, Nylander G, Kvist J. Hand function and quality of life before and after fasciectomy for Dupuytren contracture. J Hand Surg Am. 2014 Jul;39(7):1333-1343.e2. doi: 10.1016/j.jhsa.2014.04.029. PMID 24969497
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Background] Mojallal A, Lequeux C, Shipkov C, Breton P, Foyatier JL, Braye F, Damour O. Improvement of skin quality after fat grafting: clinical observation and an animal study. Plast Reconstr Surg. 2009 Sep;124(3):765-774. doi: 10.1097/PRS.0b013e3181b17b8f. PMID 19730294
- [Background] Verhoekx JSN, Mudera V, Walbeehm ET, Hovius SER. Adipose-derived stem cells inhibit the contractile myofibroblast in Dupuytren's disease. Plast Reconstr Surg. 2013 Nov;132(5):1139-1148. doi: 10.1097/PRS.0b013e3182a3bf2b. PMID 23924646
- [Background] Foucher G, Medina J, Navarro R. Percutaneous needle aponeurotomy: complications and results. J Hand Surg Br. 2003 Oct;28(5):427-31. doi: 10.1016/s0266-7681(03)00013-5. PMID 12954251
- [Background] Kan HJ, Verrijp FW, Hovius SER, van Nieuwenhoven CA; Dupuytren Delphi Group; Selles RW. Recurrence of Dupuytren's contracture: A consensus-based definition. PLoS One. 2017 May 15;12(5):e0164849. doi: 10.1371/journal.pone.0164849. eCollection 2017. PMID 28505187
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Derived] Sawaya ET, Sommier B, Alet JM, Piechaud PT; REMEDY Study Group; ReSurg; Lecoq FA. Limited fasciectomy with versus without autologous adipose tissue grafting for treatment of Dupuytren's contracture (REMEDY): study protocol for a multicentre randomised controlled trial. Trials. 2024 Sep 2;25(1):577. doi: 10.1186/s13063-024-08410-4. PMID 39223657